CLINICAL TRIAL: NCT00474318
Title: Teen-Longitudinal Assessment of Bariatric Surgery (Teen-LABS) Research Project
Brief Title: Teen-Longitudinal Assessment of Bariatric Surgery (Teen-LABS) Adolescent Bariatrics: Assessing Health Benefits and Risk
Acronym: Teen-LABS
Status: Completed | Type: Observational
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Children's Hospital Medical Center, Cincinnati (Other); University of Pittsburgh Medical Center (Other); University of Alabama at Birmingham (Other); Nationwide Children's Hospital (Other); Baylor College of Medicine (Other); Sanford Health (Other); University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 17-0235; 7UM1DK072493-17 (NIH); 5UM1DK095710-10 (NIH); 5UM1DK072493-16 (NIH)
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Obesity
Keywords: Adolescents; Obesity; Bariatrics; Surgery for Weight Loss; Teen-LABS
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma and urine, as well as liver samples (if agreed upon as part of the study; may participate in the study without giving samples per Informed Consent)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adolescents with severe obesity: Adolescents and young adults with severe obesity

SUMMARY:
The five Teen-LABS clinical centers use standardized techniques to assess the short and longer-term safety and efficacy of bariatric surgery in adolescents compared to adults.

DETAILED DESCRIPTION:
The goal of Teen-LABS is to facilitate coordinated clinical, epidemiological and behavioral research in the field of adolescent bariatric surgery, through the cooperative development of common clinical protocols and a bariatric surgery database that will collect information from participating clinical centers performing bariatric surgery on teenagers.

Teen-LABS will help pool the necessary clinical expertise and administrative resources to facilitate the conduct of multiple clinical studies in a timely, efficient manner. Also, the use of standardized definitions, shared clinical protocols and data collection instruments will enhance investigators' ability to provide meaningful evidence-based recommendations for patient evaluation, selection and follow-up care.

In addition to investigating surgical outcomes, another broader goal of Teen-LABS is to better understand the etiology, pathophysiology, and behavioral aspects of severe obesity in youth and how this condition affects human beings over time.

In the 3rd five year cycle of funding for this project, several additional long-term research aims have been added, all in general alignment with the original aims of the project to assess efficacy and safety of bariatric surgery performed in adolescent years.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents up to age 19
* Approved for bariatric surgery
* Agreement to participate in Teen-LABS Study/ understand and sign Informed Consent/Assent

Exclusion Criteria:

* Age 19 or greater
* Unable to sign Informed Consent/Assent

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents and young adults who were approved to undergo bariatriac surgery, at a participating study site, by a Teen-LABS approved surgeon, that have signed Informed Consent to participate in the study
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2007-03; Primary Completion 2024-06 (Actual); Study Completion 2024-06 (Actual)

PRIMARY OUTCOMES:
Percent change in body mass index from baseline measurement. | Calculated at each study time point following baseline (i.e., 6 months, 1 year, and annually thereafter through 10 years).
  Body mass index is calculated as kilograms divided by height in meters squared. Percent change in body mass index from baseline is calculated as: [(Follow-up BMI - Baseline BMI) /Baseline BMI]*100%.
Change in number of participants achieving remission from baseline Type II diabetes. | Determined at each study time point following baseline (i.e., 6 months, 1 year, and annually thereafter through 10 years).
  Among those subjects identified with diabetes (DM) at baseline, remission of DM at each post-operative study time point was defined as: no use of medication for DM, and HbA1c < 6.5%, or, if HbA1c was not available, fasting glucose <126mg/dL. DM at baseline was defined by taking into consideration self-report of prior diagnosis, as well as prior medical records from referring physician, use of DM medications, baseline HbA1c ≥6.5%, fasting glucose ≥126 mg/dL, or oral glucose tolerance results in prior 6 months. Participants reporting having polycystic ovarian syndrome who did not meet laboratory criteria for diabetes and were not taking a DM medication other than metformin were not considered to have DM. Participants who were on metformin at baseline for weight management or for insulin resistance, with no other indication of a prior diagnosis of DM documented and no laboratory findings consistent with the diagnosis of DM were not considered to have DM.
Change in number of participants achieving remission from baseline Hypertension. | Determined at each study time point following baseline (i.e., 6 months, 1 year, and annually thereafter through 10 years).
  Among those subjects identified with hypertension (HTN) at baseline, remission of HTN was defined as that no medications for blood pressure (BP) were being used and systolic BP < 140 mmHg and diastolic BP < 90 mmHg. BP was measured at the time of the study visit and use of medications for control of BP was recorded on medication use form (MED). Hypertension was defined in a manner consistent with that used to clinically define hypertension: use of BP medications or systolic BP>140 mmHg or diastolic BP > 90 mmHg.

SECONDARY OUTCOMES:
Number of participants with Hypoferritinemia. | Determined at each study time point (i.e., baseline, 6 months, 1 year, and annually thereafter through 10 years).
  Fasting blood specimens were drawn at the preoperative, 6 month, and annual research visits. All laboratory assays were performed by the Northwest Lipid Metabolism and Diabetes Research Laboratories (Seattle, WA). Presence of hypoferritinemia is defined as <10ug/L for females and <20ug/L for males.
Number of participants with Hypovitaminosis B12. | Determined at each study time point (i.e., baseline, 6 months, 1 year, and annually thereafter through 10 years).
  Fasting blood specimens were drawn at the preoperative, 6 month, and annual research visits. All laboratory assays were performed by the Northwest Lipid Metabolism and Diabetes Research Laboratories (Seattle, WA). Presence of hypovitaminosis B12 is defined as <145pg/mL.
Occurrence of Abdominal re-operations. | Occurrence of abdominal re-operations are identified at each study time point following baseline (i.e., 6 months, 1 year, and annually thereafter through 10 years).
  Abdominal re-operations were identified from the following data collection instruments: Discharge Summary, Post-operative Evaluation, and Healthcare Utilization forms.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Inge, MD, PhD, Study Chair — Ann & Robert H Lurie Children's Hospital of Chicago; Stephanie Sisley, MD, Principal Investigator — Baylor College of Medicine; Mike Chen, MD, Principal Investigator — University of Alabama at Birmingham; Anita P Courcoulas, MD, MPH, Principal Investigator — University of Pittsburgh Medical Center; Todd M Jenkins, PhD,MPH, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Marc Michalsky, MD, Principal Investigator — Nationwide Children's Hospital; Michael Helmrath, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Changchun Xie, PhD, Principal Investigator — University of Cincinnati; James Mitchell, MD, Principal Investigator — Sanford Health
Locations (3):
- United States (3):
  - Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Data uploaded to NIH repository and available from publications

REFERENCES:
- [Background] Chidambaran V, Venkatasubramanian R, Sadhasivam S, Esslinger H, Cox S, Diepstraten J, Fukuda T, Inge T, Knibbe CAJ, Vinks AA. Population pharmacokinetic-pharmacodynamic modeling and dosing simulation of propofol maintenance anesthesia in severely obese adolescents. Paediatr Anaesth. 2015 Sep;25(9):911-923. doi: 10.1111/pan.12684. Epub 2015 May 13. PMID 25975390
- [Background] Inge TH, Courcoulas AP, Jenkins TM, Michalsky MP, Helmrath MA, Brandt ML, Harmon CM, Zeller MH, Chen MK, Xanthakos SA, Horlick M, Buncher CR; Teen-LABS Consortium. Weight Loss and Health Status 3 Years after Bariatric Surgery in Adolescents. N Engl J Med. 2016 Jan 14;374(2):113-23. doi: 10.1056/NEJMoa1506699. Epub 2015 Nov 6. PMID 26544725
- [Background] Gowey MA, Reiter-Purtill J, Becnel J, Peugh J, Mitchell JE, Zeller MH; TeenView Study Group. Weight-related correlates of psychological dysregulation in adolescent and young adult (AYA) females with severe obesity. Appetite. 2016 Apr 1;99:211-218. doi: 10.1016/j.appet.2016.01.020. Epub 2016 Jan 14. PMID 26775646
- [Background] Xanthakos SA, Jenkins TM, Kleiner DE, Boyce TW, Mourya R, Karns R, Brandt ML, Harmon CM, Helmrath MA, Michalsky MP, Courcoulas AP, Zeller MH, Inge TH; Teen-LABS Consortium. High Prevalence of Nonalcoholic Fatty Liver Disease in Adolescents Undergoing Bariatric Surgery. Gastroenterology. 2015 Sep;149(3):623-34.e8. doi: 10.1053/j.gastro.2015.05.039. Epub 2015 May 28. PMID 26026390
- [Background] Bout-Tabaku S, Michalsky MP, Jenkins TM, Baughcum A, Zeller MH, Brandt ML, Courcoulas A, Buncher R, Helmrath M, Harmon CM, Chen MK, Inge TH. Musculoskeletal Pain, Self-reported Physical Function, and Quality of Life in the Teen-Longitudinal Assessment of Bariatric Surgery (Teen-LABS) Cohort. JAMA Pediatr. 2015 Jun;169(6):552-9. doi: 10.1001/jamapediatrics.2015.0378. PMID 25915190
- [Background] Michalsky MP, Inge TH, Simmons M, Jenkins TM, Buncher R, Helmrath M, Brandt ML, Harmon CM, Courcoulas A, Chen M, Horlick M, Daniels SR, Urbina EM; Teen-LABS Consortium. Cardiovascular Risk Factors in Severely Obese Adolescents: The Teen Longitudinal Assessment of Bariatric Surgery (Teen-LABS) Study. JAMA Pediatr. 2015 May;169(5):438-44. doi: 10.1001/jamapediatrics.2014.3690. PMID 25730293
- [Background] Zeller MH, Inge TH, Modi AC, Jenkins TM, Michalsky MP, Helmrath M, Courcoulas A, Harmon CM, Rofey D, Baughcum A, Austin H, Price K, Xanthakos SA, Brandt ML, Horlick M, Buncher R; Teen Longitudinal Assessment of Bariatric Surgery (Teen-LABS) Consortium. Severe obesity and comorbid condition impact on the weight-related quality of life of the adolescent patient. J Pediatr. 2015 Mar;166(3):651-9.e4. doi: 10.1016/j.jpeds.2014.11.022. Epub 2014 Dec 30. PMID 25556022
- [Background] Butte NF, Brandt ML, Wong WW, Liu Y, Mehta NR, Wilson TA, Adolph AL, Puyau MR, Vohra FA, Shypailo RJ, Zakeri IF. Energetic adaptations persist after bariatric surgery in severely obese adolescents. Obesity (Silver Spring). 2015 Mar;23(3):591-601. doi: 10.1002/oby.20994. PMID 25707380
- [Background] Jeffreys RM, Inge TH, Jenkins TM, King WC, Oruc V, Douglas AD, Bray MS. Physical activity monitoring in extremely obese adolescents from the Teen-LABORATORIES study. J Phys Act Health. 2015 Jan;12(1):132-8. doi: 10.1123/jpah.2013-0006. Epub 2014 Sep 10. PMID 25205688
- [Background] Xiao N, Jenkins TM, Nehus E, Inge TH, Michalsky MP, Harmon CM, Helmrath MA, Brandt ML, Courcoulas A, Moxey-Mims M, Mitsnefes MM; Teen-LABS Consortium. Kidney function in severely obese adolescents undergoing bariatric surgery. Obesity (Silver Spring). 2014 Nov;22(11):2319-25. doi: 10.1002/oby.20870. PMID 25376399
- [Background] Inge TH, Zeller M, Harmon C, Helmrath M, Bean J, Modi A, Horlick M, Kalra M, Xanthakos S, Miller R, Akers R, Courcoulas A. Teen-Longitudinal Assessment of Bariatric Surgery: methodological features of the first prospective multicenter study of adolescent bariatric surgery. J Pediatr Surg. 2007 Nov;42(11):1969-71. doi: 10.1016/j.jpedsurg.2007.08.010. No abstract available. PMID 18022459
- [Background] Inge TH, Zeller MH, Jenkins TM, Helmrath M, Brandt ML, Michalsky MP, Harmon CM, Courcoulas A, Horlick M, Xanthakos SA, Dolan L, Mitsnefes M, Barnett SJ, Buncher R; Teen-LABS Consortium. Perioperative outcomes of adolescents undergoing bariatric surgery: the Teen-Longitudinal Assessment of Bariatric Surgery (Teen-LABS) study. JAMA Pediatr. 2014 Jan;168(1):47-53. doi: 10.1001/jamapediatrics.2013.4296. PMID 24189578
- [Background] Hillman JB, Miller RJ, Inge TH. Menstrual concerns and intrauterine contraception among adolescent bariatric surgery patients. J Womens Health (Larchmt). 2011 Apr;20(4):533-8. doi: 10.1089/jwh.2010.2462. Epub 2011 Mar 17. PMID 21413894
- [Background] Modi AC, Zeller MH, Xanthakos SA, Jenkins TM, Inge TH. Adherence to vitamin supplementation following adolescent bariatric surgery. Obesity (Silver Spring). 2013 Mar;21(3):E190-5. doi: 10.1002/oby.20031. PMID 23404956
- [Background] Sawhney P, Modi AC, Jenkins TM, Zeller MH, Kollar LM, Inge TH, Xanthakos SA. Predictors and outcomes of adolescent bariatric support group attendance. Surg Obes Relat Dis. 2013 Sep-Oct;9(5):773-9. doi: 10.1016/j.soard.2013.03.016. Epub 2013 May 3. PMID 23810608
- [Background] Jenkins TM, Wilson Boyce T, Akers R, Andringa J, Liu Y, Miller R, Powers C, Ralph Buncher C. Evaluation of a Teleform-based data collection system: a multi-center obesity research case study. Comput Biol Med. 2014 Jun;49:15-8. doi: 10.1016/j.compbiomed.2014.03.002. Epub 2014 Mar 13. PMID 24709056
- [Background] Michalsky MP, Raman SV, Teich S, Schuster DP, Bauer JA. Cardiovascular recovery following bariatric surgery in extremely obese adolescents: preliminary results using Cardiac Magnetic Resonance (CMR) Imaging. J Pediatr Surg. 2013 Jan;48(1):170-7. doi: 10.1016/j.jpedsurg.2012.10.032. PMID 23331811
- [Background] Chuang J, Zeller MH, Inge T, Crimmins N. Bariatric surgery for severe obesity in two adolescents with type 1 diabetes. Pediatrics. 2013 Oct;132(4):e1031-4. doi: 10.1542/peds.2012-3640. Epub 2013 Sep 23. PMID 24062368
- [Background] Kaulfers AM, Bean JA, Inge TH, Dolan LM, Kalkwarf HJ. Bone loss in adolescents after bariatric surgery. Pediatrics. 2011 Apr;127(4):e956-61. doi: 10.1542/peds.2010-0785. Epub 2011 Mar 28. PMID 21444596
- [Background] Inge TH, King WC, Jenkins TM, Courcoulas AP, Mitsnefes M, Flum DR, Wolfe BM, Pomp A, Dakin GF, Khandelwal S, Zeller MH, Horlick M, Pender JR, Chen JY, Daniels SR. The effect of obesity in adolescence on adult health status. Pediatrics. 2013 Dec;132(6):1098-104. doi: 10.1542/peds.2013-2185. Epub 2013 Nov 18. PMID 24249816
- [Background] Michalsky MP, Inge TH, Teich S, Eneli I, Miller R, Brandt ML, Helmrath M, Harmon CM, Zeller MH, Jenkins TM, Courcoulas A, Buncher RC; Teen-LABS Consortium. Adolescent bariatric surgery program characteristics: the Teen Longitudinal Assessment of Bariatric Surgery (Teen-LABS) study experience. Semin Pediatr Surg. 2014 Feb;23(1):5-10. doi: 10.1053/j.sempedsurg.2013.10.020. Epub 2013 Oct 31. PMID 24491361
- [Background] Lokken KL, Boeka AG, Austin HM, Gunstad J, Harmon CM. Evidence of executive dysfunction in extremely obese adolescents: a pilot study. Surg Obes Relat Dis. 2009 Sep-Oct;5(5):547-52. doi: 10.1016/j.soard.2009.05.008. Epub 2009 Jun 23. PMID 19766958
- [Background] Diepstraten J, Chidambaran V, Sadhasivam S, Esslinger HR, Cox SL, Inge TH, Knibbe CA, Vinks AA. Propofol clearance in morbidly obese children and adolescents: influence of age and body size. Clin Pharmacokinet. 2012 Aug 1;51(8):543-51. doi: 10.2165/11632940-000000000-00000. PMID 22690673
- [Background] Chidambaran V, Sadhasivam S, Diepstraten J, Esslinger H, Cox S, Schnell BM, Samuels P, Inge T, Vinks AA, Knibbe CA. Evaluation of propofol anesthesia in morbidly obese children and adolescents. BMC Anesthesiol. 2013 Apr 21;13:8. doi: 10.1186/1471-2253-13-8. eCollection 2013. PMID 23602008
- [Background] Diepstraten J, Chidambaran V, Sadhasivam S, Blusse van Oud-Alblas HJ, Inge T, van Ramshorst B, van Dongen EP, Vinks AA, Knibbe CA. An integrated population pharmacokinetic meta-analysis of propofol in morbidly obese and nonobese adults, adolescents, and children. CPT Pharmacometrics Syst Pharmacol. 2013 Sep 11;2(9):e73. doi: 10.1038/psp.2013.47. PMID 24026252
- [Background] Ratcliff MB, Zeller MH, Inge TH, Hrovat KB, Modi AC. Feasibility of ecological momentary assessment to characterize adolescent postoperative diet and activity patterns after weight loss surgery. Surg Obes Relat Dis. 2014 Jul-Aug;10(4):705-10. doi: 10.1016/j.soard.2014.01.034. Epub 2014 Feb 12. PMID 24837564
- [Background] Zeller MH, Noll JG, Sarwer DB, Reiter-Purtill J, Rofey DL, Baughcum AE, Peugh J, Courcoulas AP, Michalsky MP, Jenkins TM, Becnel JN; TeenView Study Group and in Cooperation With Teen-LABS Consortium. Child Maltreatment and the Adolescent Patient With Severe Obesity: Implications for Clinical Care. J Pediatr Psychol. 2015 Aug;40(7):640-8. doi: 10.1093/jpepsy/jsv011. Epub 2015 Mar 15. PMID 25774054
- [Background] Utzinger LM, Gowey MA, Zeller M, Jenkins TM, Engel SG, Rofey DL, Inge TH, Mitchell JE; Teen Longitudinal Assessment of Bariatric Surgery (Teen-LABS) Consortium. Loss of control eating and eating disorders in adolescents before bariatric surgery. Int J Eat Disord. 2016 Oct;49(10):947-952. doi: 10.1002/eat.22546. Epub 2016 May 19. PMID 27196378
- [Background] Zani A, Ford-Adams M, Ratcliff M, Bevan D, Inge TH, Desai A. Weight loss surgery improves quality of life in pediatric patients with osteogenesis imperfecta. Surg Obes Relat Dis. 2017 Jan;13(1):41-44. doi: 10.1016/j.soard.2015.11.029. Epub 2015 Dec 2. PMID 26948942
- [Background] Xiao N, Devarajan P, Inge TH, Jenkins TM, Bennett M, Mitsnefes MM. Subclinical kidney injury before and 1 year after bariatric surgery among adolescents with severe obesity. Obesity (Silver Spring). 2015 Jun;23(6):1234-8. doi: 10.1002/oby.21070. Epub 2015 May 9. PMID 25959555
- [Background] Rofey DL, Zeller MH, Brode C, Reiter-Purtill J, Mikhail C, Washington G, Baughcum AE, Peugh J, Austin H, Jenkins TM, Courcoulas AP; TeenView Writing Group in cooperation with the Teen-LABS Consortium. A multisite view of psychosocial risks in patients presenting for bariatric surgery. Obesity (Silver Spring). 2015 Jun;23(6):1218-25. doi: 10.1002/oby.21065. Epub 2015 May 9. PMID 25959437
- [Background] DeFoor WR, Asplin JR, Kollar L, Jackson E, Jenkins T, Schulte M, Inge T. Prospective evaluation of urinary metabolic indices in severely obese adolescents after weight loss surgery. Surg Obes Relat Dis. 2016 Feb;12(2):363-7. doi: 10.1016/j.soard.2015.03.013. Epub 2015 Mar 28. PMID 26077697
- [Background] Kelly AS, Ryder JR, Marlatt KL, Rudser KD, Jenkins T, Inge TH. Changes in inflammation, oxidative stress and adipokines following bariatric surgery among adolescents with severe obesity. Int J Obes (Lond). 2016 Feb;40(2):275-80. doi: 10.1038/ijo.2015.174. Epub 2015 Aug 28. PMID 26315843
- [Background] Zeller MH, Washington GA, Mitchell JE, Sarwer DB, Reiter-Purtill J, Jenkins TM, Courcoulas AP, Peugh JL, Michalsky MP, Inge TH; Teen-LABS Consortium and in collaboration with the TeenView Study Group. Alcohol use risk in adolescents 2 years after bariatric surgery. Surg Obes Relat Dis. 2017 Jan;13(1):85-94. doi: 10.1016/j.soard.2016.05.019. Epub 2016 May 25. PMID 27567561
- [Background] Ryder JR, Edwards NM, Gupta R, Khoury J, Jenkins TM, Bout-Tabaku S, Michalsky MP, Harmon CM, Inge TH, Kelly AS. Changes in Functional Mobility and Musculoskeletal Pain After Bariatric Surgery in Teens With Severe Obesity: Teen-Longitudinal Assessment of Bariatric Surgery (LABS) Study. JAMA Pediatr. 2016 Sep 1;170(9):871-7. doi: 10.1001/jamapediatrics.2016.1196. PMID 27429076
- [Background] Ishman S, Heubi C, Jenkins T, Michalsky M, Simakajornboon N, Inge T. OSA screening with the pediatric sleep questionnaire for adolescents undergoing bariatric surgery in teen-LABS. Obesity (Silver Spring). 2016 Nov;24(11):2392-2398. doi: 10.1002/oby.21623. Epub 2016 Sep 15. PMID 27629938
- [Background] Nehus EJ, Khoury JC, Inge TH, Xiao N, Jenkins TM, Moxey-Mims MM, Mitsnefes MM. Kidney outcomes three years after bariatric surgery in severely obese adolescents. Kidney Int. 2017 Feb;91(2):451-458. doi: 10.1016/j.kint.2016.09.031. Epub 2016 Dec 1. PMID 27914704
- [Background] Jenkins TM, Boyce TW, Ralph Buncher C, Zeller MH, Courcoulas AP, Evans M, Inge TH. Accuracy of Self-Reported Weight Among Adolescent and Young Adults Following Bariatric Surgery. Obes Surg. 2017 Jun;27(6):1529-1532. doi: 10.1007/s11695-016-2514-4. PMID 28012151
- [Background] DeFoor WR Jr, Inge TH, Jenkins TM, Jackson E, Courcoulas A, Michalsky M, Brandt M, Kollar L, Xie C. Prospective evaluation of urinary incontinence in severely obese adolescents presenting for weight loss surgery. Surg Obes Relat Dis. 2018 Feb;14(2):214-218. doi: 10.1016/j.soard.2017.09.510. Epub 2017 Sep 14. PMID 29074351
- [Background] Goldschmidt AB, Khoury J, Jenkins TM, Bond DS, Thomas JG, Utzinger LM, Zeller MH, Inge TH, Mitchell JE. Adolescent Loss-of-Control Eating and Weight Loss Maintenance After Bariatric Surgery. Pediatrics. 2018 Jan;141(1):e20171659. doi: 10.1542/peds.2017-1659. Epub 2017 Dec 13. PMID 29237801
- [Background] Michalsky MP, Inge TH, Jenkins TM, Xie C, Courcoulas A, Helmrath M, Brandt ML, Harmon CM, Chen M, Dixon JB, Urbina EM; Teen-LABS Consortium. Cardiovascular Risk Factors After Adolescent Bariatric Surgery. Pediatrics. 2018 Feb;141(2):e20172485. doi: 10.1542/peds.2017-2485. Epub 2018 Jan 8. PMID 29311357
- [Background] Inge TH, Laffel LM, Jenkins TM, Marcus MD, Leibel NI, Brandt ML, Haymond M, Urbina EM, Dolan LM, Zeitler PS; Teen-Longitudinal Assessment of Bariatric Surgery (Teen-LABS) and Treatment Options of Type 2 Diabetes in Adolescents and Youth (TODAY) Consortia. Comparison of Surgical and Medical Therapy for Type 2 Diabetes in Severely Obese Adolescents. JAMA Pediatr. 2018 May 1;172(5):452-460. doi: 10.1001/jamapediatrics.2017.5763. PMID 29532078
- [Background] Dewberry LC, Khoury JC, Ehrlich S, Jenkins TM, Beamish AJ, Kalkwarf HJ, Xanthakos SA, Inge T. Change in gastrointestinal symptoms over the first 5 years after bariatric surgery in a multicenter cohort of adolescents. J Pediatr Surg. 2019 Jun;54(6):1220-1225. doi: 10.1016/j.jpedsurg.2019.02.032. Epub 2019 Feb 28. PMID 30879757
- [Background] Inge TH, Courcoulas AP, Jenkins TM, Michalsky MP, Brandt ML, Xanthakos SA, Dixon JB, Harmon CM, Chen MK, Xie C, Evans ME, Helmrath MA; Teen-LABS Consortium. Five-Year Outcomes of Gastric Bypass in Adolescents as Compared with Adults. N Engl J Med. 2019 May 30;380(22):2136-2145. doi: 10.1056/NEJMoa1813909. Epub 2019 May 16. PMID 31116917
- [Background] Price PH, Kaizer AM, Daniels SR, Jenkins TM, Inge TH, Eckel RH. Physical Activity Improves Lipid and Weight-Loss Outcomes After Metabolic Bariatric Surgery in Adolescents with Severe Obesity. Obesity (Silver Spring). 2019 Jun;27(6):989-996. doi: 10.1002/oby.22475. Epub 2019 May 3. PMID 31050388
- [Background] Bout-Tabaku S, Gupta R, Jenkins TM, Ryder JR, Baughcum AE, Jackson RD, Inge TH, Dixon JB, Helmrath MA, Courcoulas AP, Mitchell JE, Harmon CM, Xie C, Michalsky MP; TEEN-LABS CONSORTIUM. Musculoskeletal Pain, Physical Function, and Quality of Life After Bariatric Surgery. Pediatrics. 2019 Dec;144(6):e20191399. doi: 10.1542/peds.2019-1399. Epub 2019 Nov 19. PMID 31744891
- [Background] Dewberry LC, Jalivand A, Gupta R, Jenkins TM, Beamish A, Inge TH, Courcoulas A, Helmrath M, Brandt ML, Harmon CM, Chen M, Dixon JB, Zeller M, Michalsky MP. Weight Loss and Health Status 5 Years After Adjustable Gastric Banding in Adolescents. Obes Surg. 2020 Jun;30(6):2388-2394. doi: 10.1007/s11695-020-04504-5. PMID 32124210
- [Background] Bjornstad P, Nehus E, Jenkins T, Mitsnefes M, Moxey-Mims M, Dixon JB, Inge TH. Five-year kidney outcomes of bariatric surgery differ in severely obese adolescents and adults with and without type 2 diabetes. Kidney Int. 2020 May;97(5):995-1005. doi: 10.1016/j.kint.2020.01.016. Epub 2020 Feb 3. PMID 32229096
- [Background] Brehm B, Summer S, Jenkins T, D'Alessio D, Inge T. Thermic effect of food and resting energy expenditure after sleeve gastrectomy for weight loss in adolescent females. Surg Obes Relat Dis. 2020 May;16(5):599-606. doi: 10.1016/j.soard.2020.01.025. Epub 2020 Feb 4. PMID 32146085
- [Background] Xanthakos SA, Khoury JC, Inge TH, Jenkins TM, Modi AC, Michalsky MP, Chen MK, Courcoulas AP, Harmon CM, Brandt ML, Helmrath MA, Kalkwarf HJ; Teen Longitudinal Assessment of Bariatric Surgery Consortium. Nutritional Risks in Adolescents After Bariatric Surgery. Clin Gastroenterol Hepatol. 2020 May;18(5):1070-1081.e5. doi: 10.1016/j.cgh.2019.10.048. Epub 2019 Nov 6. PMID 31706057
- [Background] Dewberry L, Khoury J, Schmiege S, Jenkins T, Boles R, Inge T. Gastrointestinal symptoms in relation to quality of life after metabolic surgery in adolescents. Surg Obes Relat Dis. 2020 Apr;16(4):554-561. doi: 10.1016/j.soard.2019.12.025. Epub 2020 Jan 3. PMID 32122816
- [Background] Zeller MH, Reiter-Purtill J, Jenkins TM, Kidwell KM, Bensman HE, Mitchell JE, Courcoulas AP, Inge TH, Ley SL, Gordon KH, Chaves EA, Washington GA, Austin HM, Rofey DL. Suicidal thoughts and behaviors in adolescents who underwent bariatric surgery. Surg Obes Relat Dis. 2020 Apr;16(4):568-580. doi: 10.1016/j.soard.2019.12.015. Epub 2019 Dec 24. PMID 32035828
- [Background] Ryder JR, Xu P, Inge TH, Xie C, Jenkins TM, Hur C, Lee M, Choi J, Michalsky MP, Kelly AS, Urbina EM. Thirty-Year Risk of Cardiovascular Disease Events in Adolescents with Severe Obesity. Obesity (Silver Spring). 2020 Mar;28(3):616-623. doi: 10.1002/oby.22725. Epub 2020 Feb 5. PMID 32090509
- [Background] Derderian SC, Patten L, Kaizer AM, Inge TH, Jenkins TM, Michalsky MP, Xie C, Dewberry LC, Sitzman TJ. Body contouring in adolescents after bariatric surgery. Surg Obes Relat Dis. 2020 Jan;16(1):137-142. doi: 10.1016/j.soard.2019.09.063. Epub 2019 Sep 18. PMID 31668945
- [Background] Bjornstad P, Hughan K, Kelsey MM, Shah AS, Lynch J, Nehus E, Mitsnefes M, Jenkins T, Xu P, Xie C, Inge T, Nadeau K. Effect of Surgical Versus Medical Therapy on Diabetic Kidney Disease Over 5 Years in Severely Obese Adolescents With Type 2 Diabetes. Diabetes Care. 2020 Jan;43(1):187-195. doi: 10.2337/dc19-0708. Epub 2019 Nov 4. PMID 31685489
- [Background] Reiter-Purtill J, Ley S, Kidwell KM, Mikhail C, Austin H, Chaves E, Rofey DL, Jenkins TM, Inge TH, Zeller MH; in cooperation with the TeenView Study Group and Teen-LABS Consortium. Change, predictors and correlates of weight- and health-related quality of life in adolescents 2-years following bariatric surgery. Int J Obes (Lond). 2020 Jul;44(7):1467-1478. doi: 10.1038/s41366-019-0394-0. Epub 2019 Jun 17. PMID 31209270
- [Background] Zeller MH, Brown JL, Reiter-Purtill J, Sarwer DB, Black L, Jenkins TM, McCracken KA, Courcoulas AP, Inge TH, Noll JG; TeenView Study Group; Teen-LABS Consortium. Sexual behaviors, risks, and sexual health outcomes for adolescent females following bariatric surgery. Surg Obes Relat Dis. 2019 Jun;15(6):969-978. doi: 10.1016/j.soard.2019.03.001. Epub 2019 Mar 20. PMID 31023575
- [Background] Rose SR, Horne VE, Bingham N, Jenkins T, Black J, Inge T. Hypothalamic Obesity: 4 Years of the International Registry of Hypothalamic Obesity Disorders. Obesity (Silver Spring). 2018 Nov;26(11):1727-1732. doi: 10.1002/oby.22315. Epub 2018 Oct 8. PMID 30296362
- [Background] Hunsaker SL, Garland BH, Rofey D, Reiter-Purtill J, Mitchell J, Courcoulas A, Jenkins TM, Zeller MH. A Multisite 2-Year Follow Up of Psychopathology Prevalence, Predictors, and Correlates Among Adolescents Who Did or Did Not Undergo Weight Loss Surgery. J Adolesc Health. 2018 Aug;63(2):142-150. doi: 10.1016/j.jadohealth.2017.12.021. Epub 2018 Apr 30. PMID 29724670
- [Background] Zeller MH, Pendery EC, Reiter-Purtill J, Hunsaker SL, Jenkins TM, Helmrath MA, Inge TH. From adolescence to young adulthood: trajectories of psychosocial health following Roux-en-Y gastric bypass. Surg Obes Relat Dis. 2017 Jul;13(7):1196-1203. doi: 10.1016/j.soard.2017.03.008. Epub 2017 Mar 22. PMID 28465159
- [Background] Sarwer DB, Dilks RJ, Spitzer JC, Berkowitz RI, Wadden TA, Moore RH, Chittams JL, Brandt ML, Chen MK, Courcoulas AP, Harmon CM, Helmrath MA, Michalsky MP, Xanthakos SA, Zeller MH, Jenkins TM, Inge TH. Changes in Dietary Intake and Eating Behavior in Adolescents After Bariatric Surgery: an Ancillary Study to the Teen-LABS Consortium. Obes Surg. 2017 Dec;27(12):3082-3091. doi: 10.1007/s11695-017-2764-9. PMID 28625002
- [Background] Reiter-Purtill J, Gowey MA, Austin H, Smith KC, Rofey DL, Jenkins TM, Garland BH, Zeller MH; TeenView Study Group and in cooperation with Teen-LABS Consortium. Peer Victimization in Adolescents With Severe Obesity: The Roles of Self-Worth and Social Support in Associations With Psychosocial Adjustment. J Pediatr Psychol. 2017 Apr 1;42(3):272-282. doi: 10.1093/jpepsy/jsw078. PMID 27680082
- [Background] Amin R, Simakajornboon N, Szczesniak R, Inge T. Early improvement in obstructive sleep apnea and increase in orexin levels after bariatric surgery in adolescents and young adults. Surg Obes Relat Dis. 2017 Jan;13(1):95-100. doi: 10.1016/j.soard.2016.05.023. Epub 2016 May 30. PMID 27720196
- [Derived] Ogle SB, Meneses EH, Kaizer AM, Moore JM, Mitchell JE, Michalsky MP, Inge T. Preoperative Weight Trends in Adolescents Undergoing Metabolic and Bariatric Surgery. Obesity (Silver Spring). 2026 Jan 29. doi: 10.1002/oby.70136. Online ahead of print. PMID 41610870
- [Derived] Baumert BO, Costello E, Li Z, Ryder JR, Inge T, Jenkins T, Sisley S, Xanthakos SA, Walker DI, Stratakis N, Valvi D, Bartell SM, Slitt AL, Kohli R, Rock S, La Merrill MA, Eckel SP, Aung MT, McConnell R, Conti DV, Chatzi L. PFAS Exposure and Postoperative Weight Regain in Adolescents After Bariatric Surgery: Findings From the Teen-LABS Study. Obesity (Silver Spring). 2025 Oct;33(10):1930-1954. doi: 10.1002/oby.70009. Epub 2025 Aug 14. PMID 40808486
- [Derived] Rode JB, Zeineddin SA, Khoury JC, Jenkins TM, Sisley SR, Courcoulas AP, Ryder JR, Michalsky MP, Inge TH. Gastroesophageal Reflux and Gastrointestinal Symptoms After Metabolic and Bariatric Surgery in Adolescents: An 8-year Follow-up Analysis. J Pediatr Surg. 2025 Apr;60(4):162215. doi: 10.1016/j.jpedsurg.2025.162215. Epub 2025 Jan 31. PMID 39933471
- [Derived] White GE, Boles RE, Courcoulas AP, Yanovski SZ, Zeller MH, Jenkins TM, Inge TH. A Prospective Cohort of Alcohol Use and Alcohol-related Problems Before and After Metabolic and Bariatric Surgery in Adolescents. Ann Surg. 2023 Sep 1;278(3):e519-e525. doi: 10.1097/SLA.0000000000005759. Epub 2022 Nov 17. PMID 36538630
- [Derived] Ogle SB, Dewberry LC, Jenkins TM, Inge TH, Kelsey M, Bruzoni M, Pratt JSA. Outcomes of Bariatric Surgery in Older Versus Younger Adolescents. Pediatrics. 2021 Mar;147(3):e2020024182. doi: 10.1542/peds.2020-024182. Epub 2021 Feb 1. PMID 33526606
- [Derived] Derderian SC, Patten L, Kaizer AM, Moore JM, Ogle S, Jenkins TM, Michalsky MP, Mitchell JE, Bjornstad P, Dixon JB, Inge TH. Influence of Weight Loss on Obesity-Associated Complications After Metabolic and Bariatric Surgery in Adolescents. Obesity (Silver Spring). 2020 Dec;28(12):2397-2404. doi: 10.1002/oby.23038. PMID 33230961